CLINICAL TRIAL: NCT06728163
Title: The Impact of Virtual Reality (VR) and Music Intervention During Preoperative Anxiety, Comprehension of Medical Explanations, and Satisfaction During Preoperative Training for Gynecology Surgical Patients Under General Anesthesia
Brief Title: Impact of Virtual Reality (VR) and Music Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 4-2023-1499
Record Dates: First submitted 2024-10-22; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: General Anesthesia
Keywords: gynecology surgical patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Written Education (Active Comparator): All procedures are conducted according to surgery protocol.Patients will receive education on the previous day before surgery, the surgery team will receive education from the previous day.The group receives written education to patients before surgery.
  Interventions: Other: written education group
- VR Educational Materials and Breathing Relaxation Language Intervention (Experimental): All procedures are carried out in accordance with the surgical protocol of Severance Hospital. Patients will receive training from the research team on the surgical procedure they will undergo on the day before the operation. The group will receive VR training materials and Verbal (non-music)-guided breathtaking instructions via VR on the day before the operation.
  Interventions: Other: VR educational material + breathing relaxation with verbal instruction
- VR Educational Materials and Breathing Relaxation Music Intervention (Experimental): All procedures are performed in accordance with the surgical protocols of Severance Hospital. Patients will receive training from the research team on the surgical procedure they will undergo on the day before the operation. The group will receive VR training materials and music-guided bridging instructions via VR on the day before the operation.
  Interventions: Other: VR educational material + breathing relaxation with music intervention
- Written Educational Materials and Breathing Relaxation Music Intervention (Experimental): All procedures are performed in accordance with the surgical protocols of Severance Hospital. Patients will receive training from the research team on the surgical procedure to be performed on the day before the operation. The group will receive written training materials and music-guided bridging instructions via VR on the day before the operation.
  Interventions: Other: written educational material + breathing relaxation with music intervention.

INTERVENTIONS:
Other: written education group — group will receive standard preoperative guidelines as common educational materials. A written notice related to surgery that was previously used in the ward is provided.
  Arms: Written Education
Other: VR educational material + breathing relaxation with verbal instruction — group will receive standard preoperative guidelines as common educational materials. The VR-based educational materials and relaxation videos will utilize custom video content developed by Film Factory. The educational content involves a visual guide, where the patient, using a VR headset, is walked through the process of entering the operating room while listening to an explanation from the operating surgeon, which takes approximately 3 minutes. Verbal instructions for breathing are provided for about 3 minutes and 3 seconds.
  Arms: VR Educational Materials and Breathing Relaxation Language Intervention
Other: VR educational material + breathing relaxation with music intervention — group will receive standard preoperative guidelines as common educational materials. The VR-based educational materials and relaxation videos will utilize custom video content developed by Film Factory. The educational content involves a visual guide, where the patient, using a VR headset, is walked through the process of entering the operating room while listening to an explanation from the operating surgeon, which takes approximately 3 minutes. The relaxation intervention, which provides instructions for calming the breath, lasts about 4 minutes and 32 seconds. After the intervention, an audio file in the form of a QR code will be provided, allowing participants to listen to it repeatedly at their discretion.
  Arms: VR Educational Materials and Breathing Relaxation Music Intervention
Other: written educational material + breathing relaxation with music intervention. — group will receive standard preoperative guidelines as common educational materials. A written notice related to surgery that was previously used in the ward is provided.
  The relaxation intervention, which provides instructions for calming the breath, lasts about 4 minutes and 32 seconds. After the intervention, an audio file in the form of a QR code will be provided, allowing participants to listen to it repeatedly at their discretion.
  Arms: Written Educational Materials and Breathing Relaxation Music Intervention

SUMMARY:
The purpose of this study is as follows.The purpose of this study is as follows. First, it aims to examine the differences in anxiety, depression, and sleep quality based on the inclusion of a music intervention during relaxation induction in the VR-based surgical education process for patients aged 20 to 65 undergoing gynecological surgery under general anesthesia. Second, it seeks to assess the impact of using virtual reality (VR) tools in preoperative education on patients' understanding of the surgical process and their satisfaction with the education.

For patients aged 20 to 65, classified as physical status 1-3 according to the American Society of Anesthesiologists (ASA) undergoing gynecological surgery under general anesthesia, educational materials related to the surgical process to be provided on the day of surgery will be created in two formats: written educational materials and virtual reality (VR) educational materials. The VR educational materials will include a relaxation-inducing breathing intervention protocol aimed at reducing anxiety. The intervention will be divided into two groups: one using verbal instructions and the other using music intervention, creating a total of four conditions.

These conditions will then be provided to the four groups, which are randomly assigned prior to surgery, to investigate whether there is a difference in preoperative anxiety, depression, and sleep quality based on the music intervention during the relaxation induction. Additionally, we aim to assess whether the provision of relaxation therapy via breathing exercises through the use of VR during the surgical education process affects patients' understanding of the surgical process and their satisfaction with the education.

DETAILED DESCRIPTION:
This study, the decision to register patients aged 20 to 65 undergoing gynecological surgery under general anesthesia will be made after obtaining consent from the patient's attending gynecologist. Patients will be informed of the study's purpose and methods in a private space, such as a consultation room in the ward or the outpatient surgery room. After at least one hour, patients who understand the study and agree to participate will be asked to provide written consent. Screening will be conducted for those who agree to participate, and patients meeting the inclusion criteria will be finally registered for the study. Double-blinding for group allocation will not be possible, and the study will proceed as a randomized prospective trial. The study coordinator (research nurse) will assign patients to the control group (written education group) and three experimental groups (VR + breathing relaxation with verbal instructions, VR + breathing relaxation with music intervention, written education + breathing relaxation with music intervention) based on a random allocation table generated using Excel. Group assignments will be made using the randomization table depending on who performs the registration.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria: Patients aged 20 to 65 undergoing gynecological surgery under general anesthesia, classified as physical status 1-3 according to the American Society of Anesthesiologists (ASA).

Exclusion Criteria:

* Patients whose surgery has been canceled
* Patients with cognitive impairment
* Patients with hearing or visual impairments
* Patients with any condition that, in the investigator's judgment, may compromise the well-being of the patient or the integrity of the study
* Individuals who are unable to read the consent form (e.g., illiterate or non-native speakers)

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 140 (Estimated)
Dates: Start 2024-03-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
K-POMS Anxiety/Depression | Baseline (pre-operative), Post-Operative Day 0 (operation day)
  K-POMS Anxiety/Depression : This scale calculates scores based on 65 items assessing six subfactors: anxiety, depression, anger, vitality, fatigue, and confusion. For the subfactors, higher scores for vitality are better, while lower scores for the negative psychological factors are better. In this study, 9 items related to anxiety and 15 items related to depression were measured using a 5-point Likert scale (4 points being "strongly agree" and 0 points being "strongly disagree").
K-RCSQ (Sleep in the ICU Questionnaire) | Baseline (pre-operative), Post-Operative Day 0 (operation day)
  K-RCSQ (Sleep in the ICU Questionnaire) : This questionnaire consists of 5 items that assess the overall quality of sleep as perceived by the patient. Each item is rated on a scale from 0 to 100, and the average score represents the quality of sleep. Higher scores indicate better sleep quality.

SECONDARY OUTCOMES:
Understanding of the Explanation : Likert | Baseline (pre-operative)
  Understanding of the explanation and educational satisfaction: These are based on a satisfaction assessment tool for web-based virtual classes developed by Im Jeong-hoon and Jeong In-seong (1999), which was modified and improved by Choi Mi-hee (2015) to evaluate the satisfaction of smartphone-based colonoscopy bowel preparation video education. Out of the 12 items in the original tool, 7 items that can be evaluated simultaneously with a written tool were used. The original tool measures aspects such as the appropriateness of educational content, methods, design, material organization, interest, and understanding, with a total of 12 items. It uses a 4-point scale (1: Not at all, 4: Very much), where higher scores indicate higher satisfaction. The reliability of the tool at the time of development was Cronbach's α = 0.84, and in Choi Mi-hee's study (2015), the reliability was Cronbach's α = 0.93. The evaluation takes approximately 3 minutes.
Educational Satisfaction : VAS | Baseline (pre-operative)
  Understanding of the explanation and educational satisfaction: These are based on a satisfaction assessment tool for web-based virtual classes developed by Im Jeong-hoon and Jeong In-seong (1999), which was modified and improved by Choi Mi-hee (2015) to evaluate the satisfaction of smartphone-based colonoscopy bowel preparation video education. Out of the 12 items in the original tool, 7 items that can be evaluated simultaneously with a written tool were used. The original tool measures aspects such as the appropriateness of educational content, methods, design, material organization, interest, and understanding, with a total of 12 items. It uses a 4-point scale (1: Not at all, 4: Very much), where higher scores indicate higher satisfaction. The reliability of the tool at the time of development was Cronbach's α = 0.84, and in Choi Mi-hee's study (2015), the reliability was Cronbach's α = 0.93. The evaluation takes approximately 3 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No